CLINICAL TRIAL: NCT07251543
Title: Effects of a Salivary Gland Massage Program on Salivary Flow , Xerostomia, Chewing, and Swallowing, and Oral Health Among Community- Dwelling Older Adults
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Chiayi Christian Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: IRB2025071
Record Dates: First submitted 2025-08-11; First posted 2025-11-26 (Actual); Last update posted 2025-11-26 (Actual); Status verified 2025-09

CONDITIONS: Oral Health Care

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Masking Description: Seed personnel
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Salivary gland massage group (Experimental): salivary gland massage
  Interventions: Behavioral: Salivary gland massage
- General oral health education group (Other): General oral health education group
  Interventions: Behavioral: General Oral Health Education

INTERVENTIONS:
Behavioral: Salivary gland massage — Participants will perform a salivary gland massage before each of their three meals, 10 times per gland, for three cycles, approximately 2 minutes each, for three months.
  Arms: Salivary gland massage group
Behavioral: General Oral Health Education — Health Education Presentation and Leaflet, Massage Not Performed
  Arms: General oral health education group

SUMMARY:
Purpose: This study aims to evaluate the effectiveness of salivary gland massage on saliva flow, xerostomia, chewing and swallowing, and oral health among community-dwelling elderly.

Design: A double-blind, randomized controlled trial, in which both participants and interventionists were unaware of group assignments.

Sample and setting: Community-dwelling older adults were recruited from community centers in Minxiong Township and were randomly assigned by center to either the intervention group (n = 54) or the control group (n = 54) using simple randomization.

Methods: the investigators conducted a randomized controlled trial with 108 older adults aged 65 and above from community centers in Chiayi County, Taiwan. Participants were randomly assigned to either an intervention group (n=54), who received guided salivary gland massage, or a control group (n=54), who received a health education leaflet on oral care. Before and after the intervention, the investigators assessed dry mouth symptoms, oral mucosal moisture, The Modified Water Swallowing Test, and Tongue Coating Index. Data were analyzed using SPSS version 22, applying chi-square tests, paired t-tests, independent t-tests, and generalized estimating equations to determine whether the massage intervention could improve saliva production, ease dry mouth, enhance chewing and swallowing functions, and promote better oral health.

Expected Research Benefits: Salivary gland massage is a simple, safe, and self-administered health promotion method. The findings of this study may serve as an intervention strategy for health promotion programs, aiming to enhance oral health and quality of life among community-dwelling older adults, while reducing the healthcare burden associated with oral health problems. Additionally, this approach may strengthen older adults' engagement in preventive health management and increase their willingness to actively manage their own health.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 65 years.
2. Mentally aware and able to express themselves in Mandarin or Taiwanese.
3. Able to follow instructions and participate in activities.
4. After the researcher explains the purpose and procedures of the study, they voluntarily participate in the study and sign the informed consent form.

Exclusion Criteria:

1. Elderly individuals with Sjögren's disease, head and neck cancer, tongue disease, or those undergoing radiation therapy or chemotherapy.
2. Those with cognitive impairment or unable to safely participate in exercise training.
3. Those unable to provide written informed consent.

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 108 (Estimated)
Dates: Start 2025-09-02 (Actual); Primary Completion 2025-12-15 (Estimated); Study Completion 2026-08-30 (Estimated)

PRIMARY OUTCOMES:
Unstimulated Salivary Flow Rate (mL/min) | 3 months
  Use 4*4 cm gauze to measure saliva. First, put the gauze into the subject's mouth and ask the subject to chew for two minutes. After two minutes, the gauze is placed in a bag, and any remaining saliva is spat into the bag and weighed. The total collected volume is recorded and converted to a flow rate per minute (mL/min). A normal baseline saliva flow rate is approximately 0.3-0.5 mL/min; a flow rate below 0.1 mL/min may indicate a risk of dry mouth.

SECONDARY OUTCOMES:
xerostomia | 3 months
  The dry mouth condition was measured using the short dry mouth questionnaire, The dry mouth questionnaire consists of 5 questions. The higher the score, the more severe the dry mouth condition.
Oral mucosal moisture measurement | 3 months
  Use an oral moisture meter to measure the wetness of the tongue dorsum mucosa. Ask the subject to stick out his tongue and measure the tongue surface 10 mm away from the tip of the tongue. Perform the measurement three times and calculate the average value.The lower the score, the more severe the dry mouth.
Swallowing assessment | 3 months
  Using a modified water swallowing test, the subject is asked to sit on a chair and swallow 5cc of water. If they can swallow smoothly, they are asked to repeat the swallowing twice and the lowest score is used as the evaluation result.A score of ≤3 indicates a failed test, signifying poor swallowing ability.
Oral health | 3 months
  Tongue coating index measurement, If Tongue coating index ≥ 50% or total score ≥ 9, oral hygiene is poor.

CONTACTS AND LOCATIONS:
Overall Officials: I-Chun Chen, AHN, Study Director — Ditmanson Medical Foundation Chia-Yi Christian Hospital
Locations (1):
- Ditmanson Medical Foundation Chiayi Christian Hospital, Chiayi City, Taiwan, Taiwan

IPD SHARING:
Plan to Share IPD: No